CLINICAL TRIAL: NCT04622176
Title: Magnetomotoric Ultrasound for Diagnostic Purposes in Rectal Cancer
Acronym: MMURC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Eva Angenete, Professor of surgery, Sahlgrenska University Hospital
Other Study IDs: MMURC
Record Dates: First submitted 2020-10-23; First posted 2020-11-09 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with rectal cancer: Patients with rectal cancer will be included and asked to participate in the study where a MMUS will be used after resection to test diagnostic accuracy.
  Interventions: Diagnostic Test: MMUS

INTERVENTIONS:
Diagnostic Test: MMUS — MMUS will be used to perform diagnostics, we will compare with MRI and histology

SUMMARY:
A magnetomotive ultrasound combines standard diagnostic ultrasound equipment with the application of an external time-varying magnetic field. The investigators aim to use this equipment to improve preoperative diagnostics in rectal cancer.

DETAILED DESCRIPTION:
The investigators will compare magnetomotive ultrasound with MRI and pathology report on specimens extracted during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Rectal cancer
* Surgery with abdominoperineal resection

Exclusion Criteria:

* No informed consent
* Not fulfilling inclusion criteria
* No rectal cancer

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with rectal cancer undergoing abdominoperineal excision.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2021-06-17 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of lymph node diagnosis compared to pathology report | 1 hour postoperatively
  Accuracy of lymph node diagnosis - a comparison between the findings with the device and the pathology report
Accuracy of lymph node diagnosis compared to MRI | 1 hour postoperatively
  Accuracy of lymph node diagnosis compared to MRI

CONTACTS AND LOCATIONS:
Overall Officials: Eva Angenete, Principal Investigator — Sahlgrenska Universitetssjukhuset
Locations (1):
- Dept. of Surgery, Sahlgrenska University Hospital/Ostra, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided